CLINICAL TRIAL: NCT01376635
Title: Depressed Cardiac Autonomic Modulation in Patients With Chronic Kidney Disease Diagnosed by Spectral Analysis of Heart Rate Variability Upon Postural Stress
Brief Title: Depressed Cardiac Autonomic Modulation in Patients With Chronic Kidney Disease Diagnosed by Spectral Analysis
Acronym: HRV
Status: Completed | Type: Observational
Sponsor: Core Educational Research and Treatment in Nephrology (Other)
Responsible Party: Carlos Alberto de Oliveira, Core Educational Research and Treatment in Nephrology
Other Study IDs: CoreEdRTNephrology
Record Dates: First submitted 2011-06-02; First posted 2011-06-20 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2008-05

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; Autonomic Dysfunction
MeSH Terms: conditions — Renal Insufficiency, Chronic; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Case-Crossover
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background/Aims: To evaluate the sympathovagal balance in patients with chronic kidney disease (CKD) on conservative treatment. Methods: In a cross-sectional study, patients with CKD stages 3, 4 and 5 not yet on dialysis (CKD group) and age-matched healthy subjects (CON group) underwent continuous heart rate recording during two twenty-minute periods in the supine position (pre-inclined), followed by passive postural inclination at 70° (inclined period). Power spectral analysis of the heart rate variability was used to assess the normalized low frequency (LFnu), indicative of sympathetic activity, and the normalized high frequency (HFnu), indicative of parasympathetic activity. The LFnu/HFnu ratio represented sympathovagal balance.

DETAILED DESCRIPTION:
Patients We evaluated 32 individuals (18 men and 14 women) with CKD at stages 3, 4 or 5 who were not yet on dialysis. The individuals were recruited at the Interdisciplinary Nucleus for Studies, Research and Treatment in Nephrology, Federal University of Juiz de Fora. All patients had been followed by a nephrologist for at least 6 months before inclusion in the study. Patients with severe cardiac disease, cancer, diabetes, collagen and demyelinating diseases, left ventricular systolic dysfunction, or a history of stroke were excluded. The control group consisted of 14 subjects with normal renal function who were non-diabetic, normotensive and free of heart disease. The study was approved by the Ethics Committee of the University Hospital of the Federal University of Juiz de Fora, document number 073/2007, and all subjects signed an informed consent before being included in the protocol.

Study Design This was a cross-sectional study in which we evaluated ANS function in patients with CKD under conservative treatment and compared the results to a control group. Power spectral analysis of the HRV at rest and during a passive orthostatic stress was performed in both groups.

Cardiovascular Evaluation The medical evaluation was performed by a cardiologist and consisted of an interview and clinical examination. Blood pressure was measured at each 2 minutes intervals using a conventional sphygmomanometer. A conventional 12-lead electrocardiogram (ECG) was performed with an electrocardiograph (model Apex 1000, TEB, Brazil). To detect LVH, we used the Cornell criterion [9]. Ventricular geometry and function were analyzed using a two-dimensional Doppler echocardiogram generated using a Philips EnVisor C Ultrasound System (Philips Medical Systems-Ultrasound, MA, USA). Measurements and indices of left ventricular function at rest were obtained through the two-dimensional and M modes, using a 3.5 MHz linear transducer placed over the third or fourth intercostal space. The diagnosis of LVH was based on the left ventricular mass index (LVMI), values for which were considered normal up to 115 g/m2 for men and up to 95 g/m2 for women [10]. The data were interpreted according to criteria established by the American Society of Echocardiography [11].

Laboratory Evaluation The results of the following tests were obtained from the patients' charts: glomerular filtration rate (eGFR; estimated from creatinine using the Modification of Diet in Renal Disease equation) [12], urea, potassium, calcium, phosphorus, hemoglobin, uric acid, parathyroid hormone (PTH), total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, glucose and urinalysis. The diagnosis of CKD was based on the Kidney Disease Outcomes Quality Initiative of the National Kidney Foundation (KDOQI/NKF) [13]: eGFR <60 ml/min/1.73 m2 and/or at least one marker of renal parenchymal damage (e.g., proteinuria), present for a period of ≥3 months.

Analysis of Heart Rate Variability The HRV was measured at rest in the supine position and during orthostatic stress. All subjects were instructed to fast for six hours and not to smoke or drink caffeine for 12 hours prior to the test. All medications that could potentially interfere with the cardiovascular response such as non-dihydropyridine calcium channel blockers, beta-blockers, central sympatholytic, tricyclic antidepressants as well as anti-arrhythmic drugs were withdrawn for at least five drug half-lives before the study. The evaluation was conducted in the morning in a calm environment with low light on a tilting table with seat belts and a platform for a footrest. The subjects underwent continuous HR recording using a Holter system (Cardio Light, Brazil) during two 20 minute periods in the supine position (pre-inclined), followed by passive postural inclination at 70° (inclined period) [14,15]. To evaluate the spectral analysis of HRV, a fast Fourier transform was used [16], obtained by means of Holter-specific software (Cardio Smart 550, Brazil), that allows periodic signals, an average of 500 sequential R-R intervals, to be divided into various bands of frequency response: ultra-low frequency (ULF: <0.0033 Hz), very low frequency (VLF: 0.0033 to 0.04 Hz), low frequency (LF: 0.04 to 0.15 Hz), and high frequency (HF: 0.15 to 0.4 Hz). The LF and HF components were used as markers of sympathetic and parasympathetic activities, respectively, and the LF/HF ratio was used as a measure of the sympathovagal balance. To minimize the effects of changes in ULF and VLF bands, the data were normalized and the results expressed as normalized units (nu). The normalization was done by dividing the power of a given component (LF or HF) by the total power spectrum; from this result, the VLF component was subtracted, and this number was then multiplied by 100. Thus, the variables used for the HRV analysis were LFnu, HFnu and the LFnu/HFnu ratio. The data were interpreted following previously published guidelines [17]. The HRV was analyzed using the highest total power expressed in msec², which was obtained after 10 minutes in the supine position and during the first 5 minutes after tilting the table.

Statistical Analysis The variables are described as mean, standard deviation, percentage or median. The descriptive statistics and normality of the data were tested by the Kolmogorov Smirnov test. The laboratory data of the control and CKD groups at baseline were compared using an independent sample T test, Chi-square test or Mann Whitney test depending on the characteristics of the variable. Spectral analysis of heart rate variability was assessed within groups in the pre-inclined and inclined periods by Kruskal Wallis or ANOVA (with post Hoc test) for both the control group and for the CKD group divided into disease stages three, four and five. The LFnu / HFnu ratio for the control and CKD groups was compared by the Mann Whitney Test. To assess the correlation between CKD stages and biochemical variables with the LFnu/HFnu ratio, Spearman's linear correlation coefficient was used. A p value less than or equal to 0.05 was considered statistically significant. All analyses were performed using SPSS 13.0 for Windows (SPSS Inc., Chicago, USA).

ELIGIBILITY:
Inclusion Criteria:

* We evaluated 32 individuals (18 men and 14 women) with CKD at stages 3, 4 or 5 who were not yet on dialysis

Exclusion Criteria:

* Patients with severe cardiac disease, cancer, diabetes, collagen and demyelinating diseases, left ventricular systolic dysfunction, or a history of stroke were excluded

Ages: 44 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with CKD stages 3, 4 and 5 not yet on dialysis (CKD group) and age-matched healthy subjects (CON group)
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2008-05; Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliveira A Carlos, MD, Principal Investigator — Core Educational Research and Treatment in Nephrology